CLINICAL TRIAL: NCT02389465
Title: Stress and Inflammation in the Pathophysiology of Late Life Depression
Brief Title: Stress and Inflammation in Late-Life Depression
Acronym: S&I
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5R01MH098260-02 (NIH)
Record Dates: First submitted 2015-02-27; First posted 2015-03-17 (Estimated); Results first posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Depression; Inflammation
Keywords: Depression; Geriatric; Inflammation
MeSH Terms: conditions — Depression; Inflammation | interventions — Escitalopram; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): This arm is for participants who are not depressed.
- Experimental - treatment (Experimental): Depressed participants will receive an antidepressant (escitalopram) AND either a non-steroidal anti-inflammatory drug (celecoxib) OR placebo (sugar pill) for 6 weeks.
  Interventions: Drug: Escitalopram + Celecoxib; Drug: Escitalopram + Placebo

INTERVENTIONS:
Drug: Escitalopram + Celecoxib — Participants will receive celecoxib in addition to escitalopram
  Arms: Experimental - treatment
Drug: Escitalopram + Placebo — Participants will receive a placebo in addition to escitalopram.
  Arms: Experimental - treatment

SUMMARY:
Over 18% of Americans aged 65 years and older have depression. Recent evidence suggests that there is a link between depression and inflammatory disease. This study investigates the relationship between inflammation in the brain and depression. Comparing biological and psychological differences in depressed and non-depressed people allows researchers to find better ways to treat and prevent depression. All participants will have: neuropsychological tests, an EKG, a spinal tap, a blood draw, and, if depressed, given either an antidepressant coupled with an anti-inflammatory medication or an anti-depressant coupled with a placebo for six weeks. The investigators are trying to correlate brain function with depression levels and biomarkers from the blood and spinal fluid.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80, male or female, any race;
2. Absence of clinical dementia
3. English speaking
4. Blood pressure not exceeding 150/90 mmHg, treated or untreated
5. Weight greater than 110 lbs
6. Normal result on liver-function test
7. No history of ulcer disease or GI bleeding
8. No renal insufficiency

Additional Inclusion Criteria for Depressed Participants:

1. DSM-IV criteria for Major Depressive Disorder
2. HAM-D greater than 18

Exclusion Criteria:

1. Known history of relevant severe drug allergy or hypersensitivity (e.g. to Citalopram or Escitalopram, and/or to celecoxib, aspirin, or other NSAIDs only for Phase 2; known demonstration of allergic-type reactions to sulfonamides);
2. Does not speak English;
3. Cannot give informed consent;
4. MRI contraindications (e.g., foreign metallic implants, pacemaker);
5. Known primary neurological disorders, such as Parkinson's disease, Alzheimer's disease, traumatic brain injury, cognitive impairment or dementia,
6. Known severe inflammatory disease such as systemic lupus erythematosis, known autoimmune diseases, such as multiple sclerosis, rheumatoid arthritis; Screen + for RF, ANA, HIV, Hepatitis B or C.
7. Clinical Dementia Rating Scale score greater than 0;
8. Diagnosis of a chronic psychiatric illness other than MDD at the discretion of the study doctor;
9. Significant handicaps (e.g. uncorrected hearing or visual impairment, mental retardation) that would interfere with testing;
10. Bleeding diathesis;
11. Severe Medical problem, which in the opinion of the investigator would pose a safety risk to the subject;
12. Clinically significant cardiovascular disease that will be assessed on a case-by-case basis. Clinically significant cardiovascular disease usually includes one or more of the following: cardiac surgery or myocardial infarction within the last 4 weeks; unstable angina; acute decompensated congestive heart failure or class IV heart failure; current significant cardiac arrhythmia or conduction disturbance, particularly those resulting in ventricular fibrillation, or causing syncope or near syncope; uncontrolled high blood pressure; QTc greater than 450msec (by history for subjects with cardiac disease); documented prior stroke;
13. Clinically significant abnormalities on EKG. Primary AV block or Right bundle branch block are not necessarily exclusionary;
14. Current diagnosis of cancer
15. Current diagnosis of HIV, active Hepatitis B and/or Hepatitis C
16. Use of an Investigational medicine within the past 30 days;
17. Use of Coumadin, Warfarin within the past 2 months;
18. Current treatment with psychotropic drugs or drugs that affect the CNS such as beta-blockers, mood stabilizers, antipsychotics, steroids or non-steroidal anti-inflammatory medications or other antidepressants. No subjects will be included in the study unless they have been off all psychotropics for at least 3 weeks, except in the case of fluoxetine, where 5 weeks off treatment will be required;
19. Current alcohol or substance abuse disorder, schizophrenia or other psychotic disorder, bipolar disorder, or current OCD;
20. Abnormal liver-function test
21. History of ulcer disease, Chron's disease, GI bleeding or anemia
22. Weight less than 110 lbs
23. Renal insufficiency
24. Any other factor that in the investigator's judgment may affect patient safety or compliance (e.g. distance greater than 100 miles from this facility);

Additional Exclusion Criteria for Depressed Subjects:

1) Active suicidality or current suicidal risk as determined by the investigator

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2014-08; Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvette Sheline, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Luning Prak ET, Brooks T, Makhoul W, Beer JC, Zhao L, Girelli T, Skarke C, Sheline YI. No increase in inflammation in late-life major depression screened to exclude physical illness. Transl Psychiatry. 2022 Mar 24;12(1):118. doi: 10.1038/s41398-022-01883-4. PMID 35332134

RESULTS

PARTICIPANT FLOW:
Recruitment Details: SEPTA and PATCO advertisements, radio advertisements on WHYY, WMGK, and WURD, Newspaper advertisements in Metro, Milestones, Golden Times, and Haddonfield Sun, recruitment flyers, iConnect, emailing doctors for referrals, and advertising in clinics
Pre-assignment Details: Total recruitment was 119 but 24 screen failed so the actual recruitment was 95
Groups:
- Healthy Control: Participants do not meet DSM-IV criteria for MDD, and did not receive any medication throughout the study
- Experimental - Placebo: Participants meet DSM-IV criteria for MDD, and received placebo pills for the 6 week duration of the study
- Escitalopram: Participants meet DSM-IV criteria for MDD and received a dose of escitalopram between 10-20mg, or a 10-20mg dose of escitalopram as well as a placebo pill daily for the 6 week duration of the study.
- Escitalopram + Celecoxib: Participants meet DSM-IV criteria for MDD and received a 10-20mg dose of escitalopram and a 400mg dose of celecoxib daily for the 6 week duration of the study
Period: Overall Study
Arm/Group | Healthy Control | Experimental - Placebo | Escitalopram | Escitalopram + Celecoxib
Started | 30 | 20 | 29 | 16
Completed | 29 | 16 | 24 | 13
Not Completed | 1 | 4 | 5 | 3
Not completed — Lost to Follow-up | 1 | 3 | 3 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants meet DSM-IV criteria for MDD, and received placebo pills for the 6 week duration of the study
- Total: Total of all reporting groups
Arm/Group | Healthy Control | Placebo | Escitalopram | Escitalopram + Celecoxib | Total
Number analyzed (Participants) | 30 | 20 | 29 | 16 | 95
Age, Customized [Count of Participants; unit: Participants]
  18-55 | 10 | 3 | 8 | 5 | 26
  56-65 | 7 | 11 | 13 | 11 | 42
  66-75 | 10 | 5 | 7 | 0 | 22
  Over 75 | 3 | 1 | 1 | 0 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 13 | 9 | 44
  Male | 17 | 11 | 16 | 7 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 29 | 20 | 28 | 16 | 93
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 11 | 10 | 14 | 5 | 40
  White | 18 | 10 | 15 | 11 | 54
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Montgomery Asberg Depression Rating Scale (MADRS) [Mean (Standard Deviation); unit: Total score (sum of points)] — This depression rating scale will be used to determine clinical outcome for depressed participants.
  Scores range from 0-60. The higher the score, the worse the outcome (see below)
  Normal: 0-6 Mild Depression: 7-19 Moderate Depression: 20-34 Severe Depression: 35+ Very Severe Depression: 60
  Total score (sum of points) | 1.27 (1.64) | 25.53 (5.41) | 27.08 (5.56) | 26.21 (4.79) | 20.02 (1.84)
IL-6 Levels [Mean (Standard Deviation); unit: pg/mL] | 4.89 (3.75) | 13.9 (10.53) | 4.12 (4.05) | 9.18 (10.29) | 8.02 (4.57)
IL-10 Levels [Mean (Standard Deviation); unit: pg/mL] | 4.8 (7.64) | 43.53 (67.4) | 13.93 (39.18) | 17.9 (27.49) | 20.04 (24.98)

OUTCOME MEASURES:

1. Primary Outcome: IL-6 Levels
Description: IL6 levels were measured in participants by blood draw 6 weeks after the first dose was given.
Time Frame: up to week 6
Population: Not everybody completed the final blood draw
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Healthy Control | Placebo | Escitalopram | Escitalopram + Celecoxib
Number analyzed (Participants) | 18 | 10 | 18 | 12
pg/mL | 5.25 (4.12) | 18.24 (15.63) | 3.69 (3.73) | 6.84 (4.83)
Statistical Analysis 1: Comparison: Healthy Control; IL6 levels in healthy controls pre- and post-treatment compared using a paired t-test; Test type: Other; p = .44, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo; IL6 levels in the placebo group pre- and post-treatment compared using a paired t-test; Test type: Other; p = .11, t-test, 2 sided
Statistical Analysis 3: Comparison: Escitalopram; IL6 levels in the escitalopram group pre- and post-treatment compared using a paired t-test; Test type: Other; p = .42, t-test, 2 sided
Statistical Analysis 4: Comparison: Escitalopram + Celecoxib; IL-6 levels in the escitalopram + celecoxib group pre- and post-treatment compared using a paired t-tes; Test type: Other; p = .49, t-test, 2 sided
Statistical Analysis 5: Comparison: Healthy Control vs Placebo vs Escitalopram vs Escitalopram + Celecoxib; IL6 levels at completion of study compared between all MDD groups (placebo, escitalopram, and escitalopram + celecoxib) and the healthy control group; Test type: Other; p = .23, t-test, 2 sided

2. Primary Outcome: Montgomery Asberg Depression Rating Scale (MADRS)
Description: This depression rating scale will be used to determine clinical outcome for depressed participants.
  Scores range from 0-60. The higher the score, the worse the outcome (see below)
  Normal: 0-6 Mild Depression: 7-19 Moderate Depression: 20-34 Severe Depression: 35+ Very Severe Depression: 60
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: Total Score (Sum of Points)
Arm/Group | Healthy Control | Placebo | Escitalopram | Escitalopram + Celecoxib
Number analyzed (Participants) | 23 | 12 | 23 | 12
Total Score (Sum of Points) | 1.27 (1.64) | 19.14 (7.92) | 14.04 (9.13) | 12.93 (9.59)
Statistical Analysis 1: Comparison: Healthy Control vs Escitalopram + Celecoxib; MADRS scores at the final visit compared between the healthy control and escitalopram + celecoxib groups; Test type: Superiority; p = .003, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Healthy Control vs Escitalopram; MADRS scores at the final visit compared between the healthy control and escitalopram groups; Test type: Superiority; p < .001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Healthy Control vs Placebo; MADRS scores at the final visit compared between the healthy control and placebo groups; Test type: Superiority; p = .034, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Placebo vs Escitalopram vs Escitalopram + Celecoxib; MADRS scores at the final visit compared between the placebo groups and all groups receiving escitalopram (both with and without celecoxib); Test type: Superiority; p = .03, ANCOVA

3. Primary Outcome: IL10 Levels
Description: IL10 levels were measured in participants by blood draw 6 weeks after the first dose was given
Time Frame: up to 6 weeks
Population: Not everybody completed the last blood draw
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Healthy Control | Placebo | Escitalopram | Escitalopram + Celecoxib
Number analyzed (Participants) | 18 | 10 | 18 | 12
pg/mL | 4.21 (5.83) | 64.9 (82.16) | 12.24 (29.32) | 18.56 (28.9)
Statistical Analysis 1: Comparison: Healthy Control; IL10 levels in healthy controls pre- and post-treatment compared using a paired t-test; Test type: Other; p = .29, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo; IL10 levels in the placebo group pre- and post-treatment compared using a paired t-test; Test type: Other; p = .19, t-test, 2 sided
Statistical Analysis 3: Comparison: Escitalopram; IL10 levels in the escitalopram group pre- and post-treatment compared using a paired t-test; Test type: Other; p = .5, t-test, 2 sided
Statistical Analysis 4: Comparison: Escitalopram + Celecoxib; IL10 levels in the escitalopram + celecoxib group pre- and post-treatment compared using a paired t-test; Test type: Other; p = .55, t-test, 2 sided
Statistical Analysis 5: Comparison: Healthy Control vs Placebo vs Escitalopram vs Escitalopram + Celecoxib; IL10 levels at completion of study compared between all MDD groups (placebo, escitalopram, and escitalopram + celecoxib) and the healthy control group; Test type: Other; p = .06, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Baseline to 6 weeks
Groups:
- Placebo: Participants meet DSM-IV criteria for MDD, and receieved placebo pills daily for the 6 week duration of the study
  Escitalopram + Placebo: Participants will receive a placebo in addition to escitalopram.
Arm/Group | Healthy Control | Placebo | Escitalopram | Escitalopram + Celecoxib
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/20 | 0/29 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/20 | 2/29 | 2/16
Other Adverse Events (participants affected / at risk) | 0/30 | 1/20 | 7/29 | 9/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Control (N=30) | Placebo (N=20) | Escitalopram (N=29) | Escitalopram + Celecoxib (N=16)
Elevated Blood Pressure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thoughts of Suicide in Response to Cognitive Task Item (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Control (N=30) | Placebo (N=20) | Escitalopram (N=29) | Escitalopram + Celecoxib (N=16)
Vasovagal Response (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 0 (0) | 4 (5) | 1 (1)
Dizziness/Light Headed (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Jittery (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinating Frequently (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Yawning Frequently (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Claustophobia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Loss of Libido (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Skin Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Grinding Teeth (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
More Tired/Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dry Mouth (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Withdraw Symptoms from Discontinuing Escitalopram Improperly (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Elevated Blood Pressure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Slipped on Escalator When Leaving Visit (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sore Chest (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sore Lower Back (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Change in Sleep Pattern (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sexual Side Effect Delayed Ejaculation (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-19): https://cdn.clinicaltrials.gov/large-docs/65/NCT02389465/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT02389465/ICF_001.pdf